CLINICAL TRIAL: NCT07084844
Title: Patient Reported Outcomes and Satisfaction With Wavelight Plus LASIK
Brief Title: Patient Reported Outcomes With WaveLight Plus LASIK
Status: Recruiting | Type: Observational
Sponsor: Mann Eye Institute (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: PB-25-02
Record Dates: First submitted 2025-07-23; First posted 2025-07-25 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism | interventions — Keratomileusis, Laser In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: WaveLigh Plus LASIK — Wavelight plus LASIK is an advanced laser eye surgery technology designed to enhance visual outcomes through personalized treatment plans. This system integrates comprehensive diagnostics, including biometry, tomography, and wavefront measurements, to create a tailored ablation profile for each patient.

SUMMARY:
This study is a single-site, single-arm, prospective, observational study of subject satisfaction, quality of vision, and quality of life after bilateral LASIK surgery. Subjects will be assessed up to 3 months post-operatively. Clinical evaluations will include refractive outcomes, visual acuity, and administration of the adapted PROWL and the Quality-of-Life Impact of Refractive Correction (QIRC) Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 39
* Meet the standard care requirements for LASIK
* Spherical equivalent (SE) more than -1.00D and up to -9.00 diopters
* Myopia ≤ -8.00 sphere (in minus cylinder format) and up to -3.00D astigmatism
* SE difference between the manifest refraction and the Sightmap measured SE being less than 0.75D
* Minimum residual stromal bed thickness of 250 µm
* If currently wearing contact lenses:

  * Soft CTL wearers discontinue for minimum 3 days
  * RGP CTL wearers discontinue for 1 month per decade of wear
* Stable refraction (2 consecutive manifest refractions within 0.25 SE)
* Stable K readings (2 consecutive K readings in 2 consecutive visits)
* Willing and able to complete all post-operative visits
* Pre-surgery BCDVA of 20/20 (0.00 logMAR) or better in each eye.Mesopic pupil size ≥ 4.5mm

Exclusion Criteria:

* Subjects with any prior ocular surgery
* Subjects with topographic evidence of keratoconus, or ectasia
* Subjects with autoimmune diseases
* Subjects who are pregnant or nursing
* Systemic disease likely to affect wound healing, such as diabetes and severe atopy
* Any ocular disease (including un-controlled dry eye) which in the investigator's opinion would affect the outcome of refractive surgery

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Eligible test subjects will be 18 to 39 years of age and who are candidates for Wavelight Plus LASIK to correct myopia or myopic astigmatism.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-09-05 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Mean score of satisfaction with uncorrected vision after wavelight plus LASIK based on PROWL-SS Questionnaire preoperative vs postoperative (question #1 [Q1] only). | 3 months postoperative

SECONDARY OUTCOMES:
PROWL-SS Questionnaire | 3 months postoperative
  PROWL-SS can be used to assess satisfaction with vision and the existence, bothersomeness and impact on usual activities in the last 7 days of four visual symptoms - double images (8 items), glare (8 items), halos (8 items) and starbursts (8 items). Subjects select one of 6 responses for each question. Responses are scaled from 0 to 100, with 0 being a worse overall outcome and 100 being a better overall outcome for the existence, bothersomeness and impact on usual activities in the last 7 days of four visual symptoms - double images (8 items), glare (8 items), halos (8 items) and starbursts (8 items).
OSDI Score | 3 months postoperative
  The OSDI© is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease. The OSDI© is a valid and reliable instrument for measuring dry eye disease (normal, mild to moderate, and severe) and effect on vision-related function.
Uncorrected distance visual acuity | 3 months postoperative
  % of eyes in each level of uncorrected visual acuity (e.g. 20/20, 20/16, 20/12.5, 20/10 with logMAR chart).

OTHER OUTCOMES:
Quality-of-Life Impact of Refractive Correction (QIRC) Questionnaire | 3 months postoperative
  QIRC can be used to measure the quality of life of people who require an optical correction (spectacles, contact lenses or refractive surgery). Subjects select one of 6 responses for each question (20 questions total). Responses are scaled from 0 to 100, with 0 being a worse overall outcome and 100 being a better overall outcome.
Manifest Refraction Spherical Equivalent | 3 months postoperative
  Percentage of eyes with post-op spherical equivalent within +/- 0.25D, 0.50D, and 0.75D respectively.
Cylinder | 3 months postoperative
  Percentage of eyes with post-op cylinder within +/- 0.25D, 0.50D, and 0.75D respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip Brunson, Principal Investigator — Mann Eye Institute
Locations (1):
- Mann Eye Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No